CLINICAL TRIAL: NCT06871813
Title: Effectiveness of an Interactive Training Program on Emergency Management Competencies Among New Nurses in China: a Controlled Trial Assessing Knowledge, Skills, and Communication
Brief Title: Effectiveness of an Interactive Training Program on Emergency Management Competencies Among New Nurses in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wenzhou Central Hospital (Other)
Responsible Party: Principal Investigator, Shupei Fang, Associate Chief Nurse, Wenzhou Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2022Y094; 2023Y0749 (Other Grant/Funding Number: Wenzhou Science and Technology Bureau)
Record Dates: First submitted 2025-03-07; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Training Effectiveness; Nurse's Role
Keywords: Emergency Management, CDIO, Escape Room, Nurses, China

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- the experimental group (Experimental): the CDIO model integrated with escape room pedagogy
  Interventions: Behavioral: combined the CDIO model with escape room pedagogy
- the control group (Experimental): receiving standard training as outlined in the new nurse syllabus
  Interventions: Behavioral: combined the CDIO model with escape room pedagogy

INTERVENTIONS:
Behavioral: combined the CDIO model with escape room pedagogy — consisting of 16 hours of theoretical instruction delivered in a classroom setting during the first two months, followed by 8 hours of practical skills training in the third month. Practical training covered four core competencies: cardiopulmonary resuscitation (CPR), closed intravenous transfusion, micro-infusion pump operation, and cardiac monitoring operation. The experimental group followed the same syllabus, incorporating an innovative teaching strategy that combined the CDIO model with escape room pedagogy.

SUMMARY:
Background Effective emergency management is essential for ensuring optimal patient outcomes, with newly enrolled nurses playing a crucial role in the early detection and intervention of critical conditions. However, in China, these nurses often encounter challenges stemming from limited clinical experience, inadequate training in emergency skills, and the lack of standardized training programs tailored to the country's unique healthcare needs. Addressing these gaps through innovative training methods is critical for enhancing patient safety and the quality of care. This randomized controlled trial aims to evaluate the effectiveness of integrating the Conceive-Design-Implement-Operate (CDIO) framework with escape room pedagogy to improve the emergency management competencies of newly enrolled nurses. The anticipated findings are expected to provide evidence-based recommendations for nursing education in China and contribute to the overall enhancement of healthcare quality in the nation.

Methods This study adopts a quasi-experimental pre-test-post-test design. Participants were divided into two groups: a control group (control group, n = 85) receiving traditional lecture-based training, and an experimental group (experimental group, n = 84) undergoing the CDIO-escape room intervention. Outcomes were evaluated using theoretical exams, operational assessments, the Clinical Emergency Response Ability Questionnaire, and the Supportive Communication Scale.

DETAILED DESCRIPTION:
Training in emergency management skills is vital for ensuring that nurses are prepared to respond effectively in critical situations. These skills encompass an integration of knowledge, practical abilities, and cognitive thinking. Research consistently demonstrates that structured training programs focused on emergency management significantly enhance nurses' theoretical knowledge, practical skills, emergency response capabilities, and communication proficiency. However, newly enrolled nurses often face challenges during rescue operations due to limited clinical experience, insufficient familiarity with first aid techniques, inadequate ability to anticipate changes in patient conditions, and underdeveloped communication skills.

In response to these challenges, the National Health Commission of China issued the Training Outline for Newly Enrolled Nurses (Trial) in 2016, which guided medical units at all levels to conduct standardized training for newly enrolled nurses, particularly in emergency management skills. Traditional lecture-based learning methods ensure a standardized approach to content delivery. However, they may fall short in addressing the hands-on skills and real-world applications critical for clinical practice. In the 21st century, adopting innovative teaching and learning strategies has become essential in nursing education. Healthcare institutions are actively exploring and implementing various innovative teaching models, such as the BOPPPS teaching model, flipped classrooms, and simulation-based training. While these methods offer valuable insights, they often fall short in fostering the combination of theoretical knowledge, practical application, and adaptability required in real-world clinical scenarios. For instance, the BOPPPS model, though effective in enhancing theoretical knowledge and practical skills, may lack the flexibility needed to cultivate adaptability in dynamic clinical environments due to its structured design. Similarly, the flipped classroom approach necessitates that students independently acquire substantial theoretical knowledge before class, which can increase stress levels and hinder comprehension for some learners. Simulation-based training, while effective in replicating clinical settings, is resource-intensive and may not fully capture the unpredictability of real emergencies. These limitations pose challenges to the comprehensive implementation of such teaching models.

The CDIO (Conceive-Design-Implement-Operate) model, introduced in 2000, is a progressive educational framework originally developed for engineering education. It emphasizes hands-on, practical learning aligned with real-world tasks. In nursing education, scholars have found that the CDIO model enables learners to better master theoretical knowledge and practical skills while enhancing independent learning, first aid proficiency, and communication abilities. Another innovative approach is the escape room, an interactive educational method where participants solve a series of puzzles and riddles within a limited time to achieve a specific goal, such as escaping from a themed room. The American Association of Medical Colleges has highlighted that escape rooms can enhance students' experiential learning by providing a dynamic and interactive environment. For instance, a study used an escape room to orient paraclinical medical students to simulated medical environments, finding that it significantly improved students' confidence and preparedness for subsequent simulation activities. Similarly, another study employed an escape room in reproductive endocrinology and infertility education, concluding that it enhanced teamwork, critical thinking, and knowledge retention. Previous study explored the use of escape rooms for training acute care professionals in Crew Resource Management and teamwork, demonstrating that this method effectively improved participants' teamwork and communication skills. Collectively, these studies suggest that escape rooms can significantly enhance emergency response capabilities, communication skills, and overall learning experiences in medical education.

Despite their individual merits, existing studies have predominantly evaluated the CDIO model and escape room pedagogy in isolation, thereby neglecting their synergistic application within nurse training programs . In China, significant gaps persist in integrating these approaches, and their individual implementation is often constrained by small sample sizes and limited scope. Moreover, current research often lacks an evidence-based framework for evaluating how these methods address the unique challenges faced by newly enrolled nurses. Little attention has been given to the synergistic effects of integrating these strategies to enhance nurses' preparedness for the dynamic and unpredictable nature of clinical emergencies.

This study aims to address these gaps by investigating the combined use of the CDIO model and escape room pedagogy in standardized training programs for newly enrolled nurses. Specifically, it seeks to determine how this integrated approach can improve clinical emergency skills and communication, which contributes to the development of innovative, evidence-based training strategies that align with the demands of modern nursing education and practice, particularly for China.

ELIGIBILITY:
Inclusion Criteria:(1) an associate degree or bachelor's degree in nursing; (2) participation in standardized training as required; (3) no prior training in the emergency department; (4) a signed informed consent form.

-

Exclusion Criteria:(1) new nurses who have already completed standardized training at other hospitals; (2) those who withdraw from the study and are unable to complete the training for any reason.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Assessment Scores | Four months
  Theoretical and operational assessments were developed based on the New Nurse Training Guidelines by five nursing experts. Operational scores focused on four core procedures: cardiopulmonary resuscitation, closed intravenous transfusion, micro-infusion pump operation, and electrocardiogram monitoring. A percentage-based scoring system was used, with the final score being an average of the four procedures. Nursing experts conducting the assessments were blinded to the experimental details.

SECONDARY OUTCOMES:
Clinical Emergency Response Ability Questionnaire | Four months
  The 28-item validated questionnaire with an internal consistency of Cronbach's α coefficient of 0.93 is adopted to evaluate emergency response abilities across five dimensions: theoretical knowledge, critical care observation, first aid response, first aid handling, and emergency management. Items are scored on a 5-point Likert scale, ranging from 1 (completely inconsistent) to 5 (completely consistent), with higher scores indicating stronger emergency skills.

CONTACTS AND LOCATIONS:
Locations (1):
- Wenzhou Central Hospital, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
The original data is available upon reasonable request from the corresponding author.